CLINICAL TRIAL: NCT07385378
Title: Effects of Myofascial Chain Tension Modulation Combined With Scapular Corrective Exercise on Scapular Movement Performance and Functional Outcomes in Tennis Players With Subacromial Impingement Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH114-REC3-210
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Subacromial Impingement Syndrome
Keywords: muscle imbalance; scapular dyskinesis; instrument-assisted soft tissue mobilization
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated scapular rehabilitation training (Instrument-Assisted Soft Tissue Mobilization+ Exercise) (Experimental): The integrated scapular rehabilitation training group received a specially designed scapular core rehabilitation program, which included the use of IASTM to inhibit overactive and tight muscles, targeted stretching exercises, strengthening training for elongated or weakened muscles, and finally, movement integration through multi-joint exercises.
  Interventions: Device: Instrument-Assisted Soft Tissue Mobilization; Device: Elastic band
- Conventional rehabilitation (Stretch+ Exercise) (Active Comparator): The conventional rehabilitation training group received only traditional rehabilitation exercises, including stretching and strengthening training.
  Interventions: Device: Elastic band

INTERVENTIONS:
Device: Instrument-Assisted Soft Tissue Mobilization — IASTM is an assistive instrument designed to reduce the physical effort required by the practitioner and can be applied without a specific directional pattern. It aims to induce localized reactive hyperemia through repeated application, temporarily alter tissue rheological properties, and modulate sensory feedback via cutaneous mechanoreceptors. Its mechanisms involve both mechanical and neurophysiological components.
  Arms: Integrated scapular rehabilitation training (Instrument-Assisted Soft Tissue Mobilization+ Exercise)
Device: Elastic band — Elastic resistance bands of different colors were used for resistance training, with training intensity increased or decreased by selecting bands of varying resistance levels.

SUMMARY:
Subacromial Impingement Syndrome (SIS) is characterized by abnormal scapular motion, including decreased upward rotation, increased internal rotation, and excessive anterior tilting, which impair shoulder and arm function. Integrated scapular rehabilitation combines Instrument-Assisted Soft Tissue Mobilization (IASTM) and postural correction exercises. IASTM detects soft tissue restrictions through multidirectional strokes and enhances the pain threshold of myofascial trigger points (MTrPs) via reflex hyperemia. Postural correction exercises aim to strengthen weakened muscles and stretch tight ones to improve stability and posture. The combination of these interventions may enhance scapular stability and dynamic control. This study aimed to investigate the effects of integrated scapular rehabilitation on scapular kinematics, movement correction, functional improvement, and pain management in tennis athletes with SIS. A two-way repeated-measures ANOVA was used to analyze pre- and post-intervention effects.

DETAILED DESCRIPTION:
Participants aged 20 years or older were recruited. Outcome measures included pain intensity, Shoulder Pain and Disability Index (SPADI), shoulder range of motion (flexion, abduction, internal and external rotation), modified Scapular Assistance Test (mSAT), muscle strength (upper, middle, and lower trapezius; serratus anterior; rhomboids; levator scapulae; internal and external rotators), soft tissue elasticity (upper trapezius), myofascial trigger point pain threshold (upper trapezius, pectoralis minor, levator scapulae, rhomboids), subacromial space, and supraspinatus thickness.

ELIGIBILITY:
Inclusion Criteria:

* Participants were included if they met all of the following conditions:

  1. a VAS score greater than 3 during the Hawkins test (indicating mild to moderate pain),
  2. at least two positive results among the Hawkins test, Neer test, and painful arch test, and
  3. a positive result on the mSAT. Only participants who fulfilled all three criteria were enrolled in the study.

Exclusion Criteria:

* Participants were excluded if they had a history of clavicle, scapular, or humeral fractures; shoulder dislocation; or rotator cuff surgery; positive results on the cervical compression test, apprehension test, or drop arm test; had received corticosteroid injections within the past three months; had undergone physical therapy within the past six months; or reported a VAS score higher than 9.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain (VAS score during the Hawkins test) | Participants were assessed at time points: prior to the intervention (baseline), immediately three weeks after the intervention, and at a one-month follow-up.